CLINICAL TRIAL: NCT05448209
Title: The Effect of Walking Exercise Based on the Theory of Disturbing Symptoms in Women With Breast Cancer Receiving Paclitaxel on Peripheral Neuropathy and Arthralgia-Myalgia: A Randomized Controlled Pilot Application
Brief Title: The Effect of Walking Exercise Based on TOUS on Peripheral Neuropathy and Arthralgia-Myalgia in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Deniz Ozdemir, Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 198411013011
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Peripheral Neuropathies; Arthralgia; Myalgia
Keywords: Breast Cancer; Peripheral Neuropathies; Arthralgia; Myalgia; theory
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases; Arthralgia; Myalgia

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Intervention Group Afterwards, patients taking paclitaxel-paclitaxel-herceptin will be given a nurse-led Motivational Interview about CIPN, physical activity and regular physical activity-walking. Patients will be instructed that the goal is to beat the previous number of steps each time. If he/she has problems/shortness of breath, chest pain, palpitation complaints during walking, he/she will be told to take a break from walking and rest. The study will be conducted under the supervision of a Medical Oncology specialist throughout the study, as well as the controls of patients with ongoing symptoms. Participants will be given a pedometer for regular follow-up, its use will be explained, and it will be told to mark it on the walking tracking chart. It will be emphasized that rhythmic walking is important for the pedometer to count correctly. Motivational Interview sessions will be conducted face-to-face at the beginning, week 4 and week 8.
  Interventions: Behavioral: walking exercise
- control group (No Intervention): control group will receive standard practice

INTERVENTIONS:
Behavioral: walking exercise — Intervention Group Afterwards, patients taking paclitaxel-paclitaxel-herceptin will be given a nurse-led Motivational Interview about CIPN, physical activity and regular physical activity-walking. Patients will be instructed that the goal is to beat the previous number of steps each time. If he/she has problems/shortness of breath, chest pain, palpitation complaints during walking, he/she will be told to take a break from walking and rest. The study will be conducted under the supervision of a Medical Oncology specialist throughout the study, as well as the controls of patients with ongoing symptoms. Participants will be given a pedometer for regular follow-up, its use will be explained, and it will be told to mark it on the walking tracking chart. It will be emphasized that rhythmic walking is important for the pedometer to count correctly. Motivational Interview sessions will be conducted face-to-face at the beginning, week 4 and week 8.
  Arms: Experimental

SUMMARY:
Peripheral neuropathy from paclitaxel is a cause for concern. This situation also affects the patient, family and healthcare professionals. All health personnel are responsible for its care. With this study, it will be possible to create evidence for nursing practices and increase the quality of life by relieving symptoms.

DETAILED DESCRIPTION:
Unique value of the project: Chemotherapy Induced Peripheral Neuropathy (CIPN) is one of the most common side effects of chemotherapeutic agents. CIPN is a frequently dose-limiting neurotoxicity that causes significant deterioration in patients' quality of life. The development of chemotherapy-induced peripheral neuropathy has not been fully explained. Due to the increasing survival rates of cancer patients, paclitaxel-induced neurotoxicity has become a growing epidemiological problem. In a systematic review to identify metabolic and lifestyle risk factors for chemotherapy-induced peripheral neuropathy in patients treated with taxane and platinum; it has been shown that the overall incidence of neuropathy varies between 16.9% and 89.4%. However, growing evidence suggests that exercise may help reduce CIPN. Specifically, the most evidence supports that moderate to vigorous aerobic exercise combined with strength and/or balance training in the clinic and at home can reduce CIPN during and after chemotherapy treatment. Physical exercise can attenuate CIPN through its effect on blood circulation/oxidative stress, inflammation, neurotransmitters, endogenous opioids, growth factors, neuroplasticity and coping, symptom interaction mechanisms. Treatment with taxane-containing chemotherapy regimens is crucial to improve overall and disease-free survival in patients with early-stage invasive breast cancer. However, taxane treatment may cause pain. Although the incidence of taxane-induced pain is inconsistent in the literature, nonspecific pain has been described in 50-78% of patients receiving taxane therapy. Myalgia and/or arthralgia experienced by patients receiving taxane-based chemotherapy may result in impaired mobility secondary to limitation of joint function, and the experience of pain may affect physical function. The beginnings of nursing theories were developed to form the foundations of nursing science through the production of profession-specific knowledge. Theories consist of concepts and statements that aim to explain or categorize phenomena related to a field of knowledge. Theory of Unpleasant Symptoms (TOUS) arises from the belief that there are common points between different symptoms. This theory allows nurses to know different symptom groups so they can recommend non-pharmacological interventions to patients.

Method: The project was planned as a prospective, single-blind, randomized controlled experimental type.

Management: Motivational interviewing is an important component of the walking intervention. Specific objectives are to evaluate the impact of gait intervention with Motivational interviewing on; CIPN severity and To evaluate the effect of walking exercise alone on arthralgia-myalgia at 12 weeks compared with standard training in breast cancer patients receiving paclitaxel.

Application

* At the stage of implementation, patients receiving Paclitaxel-Paclitaxel-Herceptin chemotherapy protocol sent by the City Hospital Medical Oncology Specialist will be interviewed and the purpose of the research will be explained and written/verbal consent will be obtained. Consent will be taken in the Oncology Training Nurse room. Patients who accept the study will be evaluated in terms of inclusion and exclusion criteria.
* Personal information form, Chemotherapy-Induced Peripheral Neuropathy Assessment Tool, McGill Melzack Pain Questionnaire, Modified BORG Scale, ECOG Performance Scale will be evaluated by interview method at the beginning of the patients who accept the study.
* Afterwards, a nurse-led Motivational Interview will be held about CIPN, physical activity and regular physical activity-walking for patients taking paclitaxel-paclitaxel-herceptin. Patients will be informed about the study and their written consent will be obtained.
* They will be told to walk at a moderate intensity, usually defined as the BORG Scale of 4 to 5 perceived effort, three to five days a week to start with 10 minutes initially, then continue until they reach 30 or 60 minutes, 3 times a week. Patients will be instructed that the goal is to exceed the previous number of steps each time.
* Participants will be informed that if they feel fatigue, lethargy, balance problems, pain, palpitations throughout the day, they can do their exercise the next day.
* If he/she has trouble/shortness of breath, chest pain, palpitation complaints during walking, he/she will be told to take a break from walking and rest. The study will be conducted under the supervision of a Medical Oncology specialist throughout the study, as well as the controls of patients with ongoing symptoms.
* Participants will be given a pedometer for regular follow-up, its use will be explained and they will be told to mark it on the walking tracking chart. How to register will be explained. The initial step count will be recorded as the number of steps recorded on the first day the patient used the pedometer.
* It will be emphasized that rhythmic walking is important for the pedometer to count correctly.
* What Is Your Biggest Physical Activity Barrier? Do you forget to be physically active? For example, if a participant's biggest obstacle is forgetting to walk, the expression of intent might be: "If it's six o'clock on Saturday, then I'll walk for 10 minutes." If then the application notification form.
* Motivational Interview sessions will be conducted face-to-face at the beginning, week 4 and week 8.
* Intervention participants will be added to a Watsap group and invited to weekly group walk events with other intervention group participants.
* They will receive a weekly written motivational message and will be encouraged to join the WhatsApp discussion.

Control Group

* Patients in the control group will receive routine training given by Oncology Education Nursing.
* Personal information form, Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT), McGill Melzack Pain Questionnaire, Modified BORG Scale, ECOG Performance in the intervention and control group by a specialist nurse at week 0, week 4, week 8, and week 12 The scale will be evaluated.
* Continuously recorded step numbers in the Intervention and Control group 0.4.8. and will be evaluated for analysis, taking into account the last measurements of the 12th week.
* A special exercise prescription, namely MG-Walking intervention support, will not be provided to control group participants. Telephone follow-up (to assess adverse events) will take place. After the completion of the training, a supervised walking exercise will be offered to the participants if they wish.

Widespread effect: This study will contribute to the literature and will have a significant impact on the quality of life of many cancer patients and cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Eastern Cooperative Oncology Group (ECOG) Status 0 to 1
* Receiving Paclitaxel or Paclitaxel-Herceptin
* Patients with 12 weeks defined in the protocol will be included.

Exclusion Criteria:

* Those with open wounds and edema on their hands and feet
* Patients with diabetes mellitus and peripheral neuropathy due to autoimmune disease
* Use other complementary therapies to prevent peripheral neuropathy throughout the treatment process.
* Conditions that limit exercise such as cardiovascular, pulmonary, musculoskeletal system
* Those with psychological and communication problems

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT) | 4 weeks after the first assessment
  The first section assesses the nine main symptoms as well as their severity, the extent to which they cause emotional disruption, and the frequency of their occurrence. The first six items in this section are related to sensory symptoms, while the seventh, eighth and ninth items are related to sub-dimensions of motor symptoms. In the second part, 14 activities were evaluated and questions were asked about the effect level of these substances. The activities assessed included fine motor and general activities. To assess the symptoms listed in the first section, "Yes" was considered equal to 1 point and "No" equal to 0 (0-9); their severity, symptoms, extent and frequency of emotional impairment were scored between 0 and 10 (0-270). The total score for the first part of the instrument is between 0 and 279. The effect level on the 14 activities in the second part was calculated between 0 and 10 (0-140). The Cronbach's alpha value of the original scale is 0.95

CONTACTS AND LOCATIONS:
Overall Officials: Selda Arslan, Phd, Study Director — Necmettin Erbakan University Faculty of Nursing
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No